CLINICAL TRIAL: NCT05651997
Title: Randomized Study Comparing Two Methods for the Treatment of Large Chondral and Osteochondral Defects of the Knee: Augmented Microfracture Technique vs. 3rd Generation of ACI
Brief Title: Study Comparing Two Methods for the Treatment of Large Chondral and Osteochondral Defects of the Knee
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Lee Ann LAURENT APPLEGATE (Unknown); Virginie PHILIPPE (Unknown)
Responsible Party: Principal Investigator, Dr. Robin Martin, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMT_MACT_OTR
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Articular Cartilage Defect; Chondral Defect; Osteochondritis
Keywords: Cellular therapy; Human articular chondrocytes
MeSH Terms: conditions — Osteochondritis

STUDY DESIGN:
Intervention Model Description: Two arms: AMT and MACT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Matrix-Assisted Autologous Chondrocytes Transplantation (MACT) (Experimental): Matrix-Assisted Autologous Chondrocytes Transplantation (MACT, also called third generation of autologous chondrocyte implantation) is based on the use of type I/III collagen membrane as a three-dimensional structural support on which autologous articular chondrocytes are seeded and cultured to form cartilage prior to implantation.
  Interventions: Procedure: MACT
- The Augmented Microfracture Technique (AMT) (Active Comparator): The Augmented Microfracture Technique (AMT, also called Autologous Matrix-Induced Chondrogenesis or AMIC) which is part of a therapeutic continuum, combines a microfracture treatment with the application of a type I/III collagen membrane. The principle is to cover the microfractured area with a resorbable membrane to stabilize the formed blood clot in order to increase the concentration of mesenchymal stem cells and promote their differentiation into a repaired tissue.
  Interventions: Procedure: AMT

INTERVENTIONS:
Procedure: MACT — * A biopsy of healthy cartilage is taken from a non-weight bearing area of the knee joint during an arthroscopic procedure.
  * The biopsy is processed in the GMP accredited laboratory to isolate and amplify chondrocytes.
  * The cells are seeded and cultured on a collagen matrix (Chondro-Gide®, Geistlich Pharma)
  * The membrane is implanted and sutured onto the injured site.
  Other Names: Third generation of ACI
  Arms: Matrix-Assisted Autologous Chondrocytes Transplantation (MACT)
Procedure: AMT — This treatment combines the microfracture procedure with the application of a bilayer matrix of porcine type I/III collagen (Chondro-Gide, Geistlich Pharma) and the supplementation of autologous bone.
  Other Names: AMIC
  Arms: The Augmented Microfracture Technique (AMT)

SUMMARY:
The major objective of this study is to evaluate the efficacy of the MACT versus the AMT for the treatment of large cartilage defects in patellofemoral and femorotibial injuries.

DETAILED DESCRIPTION:
Knee cartilage injuries are common, especially in young active adults, and have the potential to progress to osteoarthritis if left untreated, which would disable a large part of the population with joint functionality loss.The issue with knee cartilage remains in the fact that the tissue has very limited healing potential as it contains no blood vessels allowing a supply in cells for a proper regeneration. Many surgical techniques have been developed for cartilage repair, however, traditional methods have shown their limitations, especially in the case of large defects. More importantly, there is no consensus on novel surgical techniques. Therefore, the choice of a proper cartilage treatment becomes crucial Worldwide, because the aging population is increasing rapidly and there is a need to remain functional and independent as long as possible.

The overall objective of the present study is to compare two advanced surgical techniques for the treatment of large defects in cartilage: one technique consists of a more conventional and widely used approach, which stimulates the natural repair of the tissue by making micro-holes in the bone, allowing the recruitment cells from the underneath bone marrow and stabilize them with a membrane to repair the defect (technique called enhanced microfracture or AMT); and the other technique called MACT, consists of taking patients own cartilage cells from a small biopsy and growing them on a membrane to form a cartilage tissue in vitro, which is then implanted surgically at the location of the injury. This second technique has the advantage of cellular assistance in the surgery enabling to improve the regeneration.

The purpose of this study is to determine which technique (AMT or MACT) is the most appropriate to treat large cartilage injuries, in order to propose the best therapeutic option depending on the severity, size and location of the injury in the joint to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 15-50 years
* Symptomatic chondral and osteochondral defect, grade III and IV according to the ICRS classification, and size between 2.5 and 15 cm2
* Failure of a conservative treatment
* Patient in good general condition, documented by an ASA score ≤ 2 (American Society of Anesthesiologists)
* Patient considered compliant and able to participate in rehabilitation and pre- and post-operative follow-up
* Consent to participate in the study

Exclusion Criteria:

* All inflammatory and synovial pathologies
* Diffuse or mirror lesions
* An unfavorable biomechanical environment
* Obesity grade II or higher, with a BMI>35 kg/m2
* Active smoking/ active drug dependency (hard drugs)
* Poor compliance
* The patient is already part of another clinical trial that may compromise the present study
* Vulnerable populations (except minors aged 15-18 years)
* Presence of open growth plate (15-18 years)
* Pregnancy or planned pregnancy during the study (MRI-related contra-indication)
* Proven allergy to penicillin and gentamicin (for MACT group) and porcine collagen (for both groups)

For final inclusion, an additional exclusion criteria will be assessed after randomization:

- Positive to HIV, HBV, HCV, syphilis.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2032-06-01 (Estimated)

PRIMARY OUTCOMES:
Patellofemoral joint-related function and quality-of-life are assessed using the Knee injury and Osteoarthritis Outcome Score (KOOS). | Change from baseline to 3, 6 12, 24, 36, 48 and 60 months post-implantation in the patellofemoral joint.
  KOOS includes five subscales: symptoms, pain, activities of daily living, function in sport/recreation, and knee-related quality of life. A score in points for each subscale will be calculated, and it ranges from 0 (worst score) to 100 (best score). Self-assessment by the patient

SECONDARY OUTCOMES:
Femorotibial joint-related function and quality-of-life are assessed using the Knee injury and Osteoarthritis Outcome Score (KOOS). | Change from baseline to 3, 6 12, 24, 36, 48 and 60 months post-implantation in the femorotibial joint.
  KOOS includes five subscales: symptoms, pain, activities of daily living, function in sport/recreation, and knee-related quality of life. A score in points for each subscale will be calculated, and it ranges from 0 (worst score) to 100 (best score).Self-assessment by the patient

OTHER OUTCOMES:
Self-reported physical pain and function are assessed by International Knee Documentation Committee score (IKDC) | Change from baseline to 3, 6 12, 24, 36, 48 and 60 months post-implantation in the patellofemoral and femorotibial joints.
  A score will be calculated, and it ranges from 0 (worst score) to 100 (best score).
Rate of implantation-associated complications: serious adverse events (SAEs) and serious adverse reactions (SARs) | Up to 60 months.
  Post-implantation data collection: Types, probability and severity of treatment (inflammation, infection,pain, joint effusion, delamination, transplant rejection, fibrocartilage, incomplete cartilage repair).
The cartilage repair is assesed by Magnetic Resonance Observation of Cartilage Repair | Change from baseline to 3, 6 12, 24, 36, 48 and 60 months post-implantation.
  MOCART scoring system is based on MRI analysis. A score in points will be calculated, and it ranges from 0 points (no repair) to 100 points (excellent cartilage defect repair)

CONTACTS AND LOCATIONS:
Overall Officials: Robin MARTIN, MD, Principal Investigator — CHUV
Locations (2):
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois - CHUV, Lausanne, Canton of Vaud
  - Hôpital Fribourgeois- HFR, Fribourg